CLINICAL TRIAL: NCT05054816
Title: Speech Locator In-car Performance Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Sonova Canada Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-459
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2021-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: A single cohort of participants will receive and be assessed in all treatment/intervention
Masking Description: Hearing aid processing settings are randomized and double blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with hearing loss. (Experimental): Participants with hearing loss.
  Interventions: Device: Investigational adaptive directional microphone strategy; Device: Comparator omnidirectional microphone strategy; Device: Comparator fixed directional microphone strategy

INTERVENTIONS:
Device: Investigational adaptive directional microphone strategy — A receiver-in-canal hearing aid developed by the Study Sponsor used with the investigational adaptive directional microphone strategy that is expected to improve sound quality of speech in a car.
Device: Comparator omnidirectional microphone strategy — A receiver-in-canal hearing aid developed by the Study Sponsor used with the comparator omnidirectional microphone strategy that is used with the default settings as specified in the manufacturer's fitting software.
Device: Comparator fixed directional microphone strategy — A receiver-in-canal hearing aid developed by the Study Sponsor used with the comparator fixed directional microphone strategy that is used with the default settings as specified in the manufacturer's fitting software.

SUMMARY:
Listeners will conduct sound quality ratings of recordings talkers in a moving car processed using three different microphone processing strategies: an investigational adaptive directional microphone, an omnidirectional microphone and a fixed directional microphone. Participants will listen to the recordings streamed via commercially-available and individually-prescribed hearing aids, and conduct ratings onsite in the lab. The procedure will involve a training session and within-subject repeated measures. Stimuli will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-99 years) with ≥3 months hearing aid experience
* binaural, symmetric, sensorineural N2 (mild) to N5 (severe) hearing loss
* fluent in English

Exclusion Criteria:

* children/teenagers
* normal hearing or hearing loss exceeding N5 (severe) by 10 dB

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova Innovation Centre Toronto, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Hearing Loss: Participants with hearing loss who are candidates for hearing aids
Period: Overall Study
Arm/Group | Participants With Hearing Loss
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Hearing Loss.
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 20
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 20
Hearing loss severity [Count of Participants; unit: Participants]
  Mild | 15
  Moderate | 3
  Moderate-Severe | 2

OUTCOME MEASURES:

1. Primary Outcome: Speech Clarity
Description: The sound quality ratings will be conducted via a computer-based questionnaire that contains sound samples that participants listen to and rate. Sound quality rating scales are continuous and range from 0 (worst) to 100 (best) with 5 descriptors unique to the dimension at 5 intervals on the scale (0, 25, 50, 75, 100)
  Participants will be instructed to "Please rate the clarity of speech". Speech clarity ratings will be measured on a 100-point continuous slider from worst to best (0-Very unclear, 25- Unclear, 50-Slightly clear, 75-Clear, 100-Very clear). Speech clarity ratings are expected to be impacted by how intelligible the speech is. Participants will rate and compare speech clarity between the investigational and comparator features.
Time Frame: Up to 6 hours over 3 2-hour sessions
Population: Two participants' data were omitted due to their results suggesting that they did not understand the task.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Participants With Hearing Loss.
Number analyzed (Participants) | 18
units on a scale
  Investigational adaptive directional microphone strategy | 77.2 (3.7)
  Comparator omnidirectional microphone strategy | 76.6 (3.7)
  Comparator fixed directional microphone strategy | 63.6 (3.7)
Statistical Analysis 1: Comparison: Participants With Hearing Loss; Previous research with subjective ratings has repeatedly shown that data collected with 15-25 participants can yield significant results; Test type: Superiority; p < 0.05, ANOVA — The p-value was adjusted for multiple comparisons between three conditions: investigative feature, comparative feature 1, comparative feature 2; The data were protected against deviations from sphericity by modifying degrees of freedom using Greenhouse-Geisser corrections

2. Primary Outcome: Noise Annoyance
Description: The sound quality ratings will be conducted via a computer-based questionnaire that contains sound samples that participants listen to and rate. Sound quality rating scales are continuous and range from 0 (worst) to 100 (best) with 5 descriptors unique to the dimension at 5 intervals on the scale (0, 25, 50, 75, 100)
  Participants will be instructed to "Please rate how annoying the noise is". Noise annoyance ratings will be measured on a 100-point continuous slider from worst to best (0- Extremely annoying, 25-Very annoying, 50-Moderately annoying, 75-Slightly annoying, 100-Not at all annoying). Noise annoyance ratings are expected to be impacted by how bothersome the background noise in the recordings is. Participants will rate and compare noise annoyance between the investigational and comparator features.
Time Frame: Up to 6 hours over 3 2-hour sessions
Population: Two participants' data were omitted due to their results suggesting that they did not understand the task.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Experimental: Participants With Hearing Loss.: Device: Investigational adaptive directional microphone strategy A receiver-in-canal hearing aid developed by the Study Sponsor used with the investigational adaptive directional microphone strategy that is expected to improve sound quality of speech in a car.
  Device: Comparator omnidirectional microphone strategy A receiver-in-canal hearing aid developed by the Study Sponsor used with the comparator omnidirectional microphone strategy that is used with the default settings as specified in the manufacturer's fitting software.
  Device: Comparator fixed directional microphone strategy A receiver-in-canal hearing aid developed by the Study Sponsor used with the comparator fixed directional microphone strategy that is used with the default settings as specified in the manufacturer's fitting software.
Arm/Group | Experimental: Participants With Hearing Loss.
Number analyzed (Participants) | 18
units on a scale
  Investigational adaptive directional microphone strategy | 71.1 (3.25)
  Comparator omnidirectional microphone strategy | 61.4 (3.25)
  Comparator fixed directional microphone strategy | 60.0 (3.25)
Statistical Analysis 1: Comparison: Experimental: Participants With Hearing Loss; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Spatialization
Description: The sound quality ratings will be conducted via a computer-based questionnaire that contains sound samples that participants listen to and rate. Sound quality rating scales are continuous and range from 0 (worst) to 100 (best) with 5 descriptors unique to the dimension at 5 intervals on the scale (0, 25, 50, 75, 100)
  Participants will be instructed to "Please rate your confidence that the talker is in [a location]", with the local being either passenger of rear left. Spatialization ratings will be measured on a 100-point continuous slider from worst to best (0-I don't know where the talker is, 25-The talker might be to my [location], 50-The talker is probably to my [location], 75-The talker is to my [location], 100-The talker is definitely to my [location]). Spatialization ratings are expected to be impacted by how well the recordings preserve spatial perception. Participants will rate and compare spatialization between the investigational and comparator features.
Time Frame: Up to 6 hours over 3 2-hour sessions
Population: Two participants' data were omitted due to their results suggesting that they did not understand the task.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Participants With Hearing Loss.
Number analyzed (Participants) | 18
units on a scale
  Investigational adaptive directional microphone strategy | 78.2 (6.42)
  Comparator omnidirectional microphone strategy | 77.7 (6.42)
  Comparator fixed directional microphone strategy | 50.5 (6.42)
Statistical Analysis 1: Comparison: Experimental: Participants With Hearing Loss; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Transition Annoyance
Description: The sound quality ratings will be conducted via a computer-based questionnaire that contains sound samples that participants listen to and rate. Sound quality rating scales are continuous and range from 0 (worst) to 100 (best) with 5 descriptors unique to the dimension at 5 intervals on the scale (0, 25, 50, 75, 100)
  Participants will be instructed to "Please rate how annoying the transitions are". Transitions annoyance ratings will be measured on a 100-point continuous slider from worst to best (0-Extremely annoying, 25-Very annoying, 50-Moderately annoying, 75-Slightly annoying, 100-Not at all annoying). Transition annoyance ratings are expected to be influenced by presence of unexpected sounds or transitions that occur in different microphone modes and different listening situations. Participants will rate and compare transition annoyance between the investigational and comparator features.
Time Frame: Up to 6 hours over 3 2-hour sessions
Population: Two participants' data were omitted due to their results suggesting that they did not understand the task. The "fixed directional" outcome measure is not included for the transition annoyance comparator since that program does not contain transitions that can be rated and compared to the other test conditions.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Participants With Hearing Loss.
Number analyzed (Participants) | 18
units on a scale
  Investigational adaptive directional microphone strategy | 71.7 (3.89)
  Comparator omnidirectional microphone strategy | 74.1 (3.89)
Statistical Analysis 1: Comparison: Experimental: Participants With Hearing Loss; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA — The p-value was adjusted for multiple comparisons between two conditions: investigative feature, comparative feature 1; [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: Overall Impression
Description: The sound quality ratings will be conducted via a computer-based questionnaire that contains sound samples that participants listen to and rate. Sound quality rating scales are continuous and range from 0 (worst) to 100 (best) with 5 descriptors unique to the dimension at 5 intervals on the scale (0, 25, 50, 75, 100)
  Participants will be instructed to "All things considered, please rate overall preferences". Overall preferences ratings will be measured on a 100-point continuous slider from worst to best (0-Bad, 25-Poor, 50-Fair, 75-Good, 100-Excellent). Overall impression ratings are expected to be impacted by participants' overall preferences for the different stimuli. Participants will rate and compare overall impression between the investigational and comparator features.
Time Frame: Up to 6 hours over 3 2-hour sessions
Population: Two participants' data were omitted due to their results suggesting that they did not understand the task.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Participants With Hearing Loss.
Number analyzed (Participants) | 18
units on a scale
  Investigational adaptive directional microphone strategy | 61 (2.8)
  Comparator omnidirectional microphone strategy | 58.7 (2.8)
  Comparator fixed directional microphone strategy | 40.6 (2.8)
Statistical Analysis 1: Comparison: Experimental: Participants With Hearing Loss; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were recorded over the course of a single 2-hour study session.
Arm/Group | Participants With Hearing Loss.
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT05054816/Prot_SAP_ICF_000.pdf